CLINICAL TRIAL: NCT00772889
Title: Safety and Immunogenicity of the Influenza Vaccine GSK2186877A in the Elderly
Brief Title: Evaluation of the Safety and Immunogenicity of the Influenza Vaccine GSK2186877A in the Elderly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 111738
Record Dates: First submitted 2008-10-10; First posted 2008-10-15 (Estimated); Results first posted 2012-04-24 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2017-04

CONDITIONS: Influenza
Keywords: Elderly; Vaccine; Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- New generation influenza vaccine GSK2186877A Group (Experimental): Subjects aged ≥66 years received one dose of New generation influenza vaccine GSK2186877A.
  Interventions: Biological: Influenza vaccine GSK2186877A
- Fluarix elderly Group (Active Comparator): Subjects aged ≥66 years received one dose of Fluarix vaccine.
  Interventions: Biological: GSK Biologicals' Fluarix™
- Fluarix young Group (Active Comparator): Subjects aged 19-43 years received one dose of Fluarix vaccine.
  Interventions: Biological: GSK Biologicals' Fluarix™

INTERVENTIONS:
Biological: Influenza vaccine GSK2186877A — One intramuscularly injection at Day 0
  Arms: New generation influenza vaccine GSK2186877A Group
Biological: GSK Biologicals' Fluarix™ — One intramuscularly injection at Day 0
  Arms: Fluarix elderly Group; Fluarix young Group

SUMMARY:
The purpose of this observer-blind clinical trial is to evaluate the safety and immunogenicity of GlaxoSmithKline Biologicals' influenza vaccine GSK2186877A in the elderly. Subjects were previously vaccinated (NCT00529516).

ELIGIBILITY:
Inclusion Criteria:

* A male or female subject previously enrolled in study 109821 (NCT 00529516) in the >= 65 years and 18-41 years of age groups and having received the study vaccine.
* Subjects of whom the investigator believes that they can and will comply with the requirements of the protocol. Specific attention should be given to the compliance potential of subjects with suspected or known drug or alcohol abuse.
* Written informed consent obtained from the subject.
* Free of an acute aggravation of the health status as established by medical history and clinical examination before entering into the study
* If the subject is female, she must be of non-childbearing potential or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Administration of other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrolment in this study.
* Planned administration of a vaccine not foreseen by the study protocol up to 30 days after vaccination.
* Planned administration of an influenza vaccine other than the study vaccines during the entire study period.
* Any vaccination against influenza since January 2008 with any seasonal influenza vaccine.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of hypersensitivity to a previous dose of influenza vaccine.
* History of allergy or reactions likely to be exacerbated by any component of the vaccines.
* Acute (active) clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or pre-existing laboratory screening tests.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the administration of the study vaccine or planned administration during the study period.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days prior to vaccination, or planned use during the study period.
* Any medical conditions in which intramuscular injections are contraindicated.
* Pregnant or lactating females.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 971 (Actual)
Dates: Start 2008-10-09; Primary Completion 2009-12-15 (Actual); Study Completion 2009-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (25):
- United States (9):
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Milford, Massachusetts
  - GSK Investigational Site, Chaska, Minnesota
  - GSK Investigational Site, Somers Point, New Jersey
  - GSK Investigational Site, Poughkeepsie, New York
  - GSK Investigational Site, Carnegie, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
- GSK Investigational Site, Ghent, Belgium
- Germany (8):
  - GSK Investigational Site, Messkirch, Baden-Wurttemberg
  - GSK Investigational Site, Augsburg, Bavaria
  - GSK Investigational Site, Haag, Bavaria
  - GSK Investigational Site, Höhenkirchen-Siegertsbrunn, Bavaria
  - GSK Investigational Site, Langquaid, Bavaria
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Berlin
- Norway (7):
  - GSK Investigational Site, Bekkestua
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Elverum
  - GSK Investigational Site, Fredrikstad
  - GSK Investigational Site, Hamar
  - GSK Investigational Site, Haugesund
  - GSK Investigational Site, Skien

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 111738 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111738 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111738 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111738 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111738 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111738 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111738 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Started | 375 | 393 | 203
Completed at Day 21 | 374 | 390 | 203
Completed | 353 | 375 | 187
Not Completed | 22 | 18 | 16
Not completed — Adverse Event | 7 | 4 | 0
Not completed — Withdrawal by Subject | 9 | 8 | 9
Not completed — Lost to Follow-up | 6 | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group | Total
Number analyzed (Participants) | 375 | 393 | 203 | 971
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74.4 (5.23) | 74.7 (5.74) | 32.4 (6.78) | 65.7 (18.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 190 | 203 | 118 | 511
  Male | 185 | 190 | 85 | 460

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Adverse Events (AEs)
Description: Grade 3 ecchymosis, redness and swelling were ≥ 100 millimeters (mm) and grade 3 pain was considerable pain at rest that prevented normal everyday activities. Any was >20 mm for ecchymosis, redness and swelling.
Time Frame: Day 0-6
Population: The analysis was performed on Total Vaccinated cohort which included all subjects with the vaccine administration documented and symptom sheet completed.
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 375 | 392 | 203
Participants
  Any ecchymosis | 2 | 3 | 1
  Grade 3 ecchymosis | 0 | 0 | 0
  Any pain | 159 | 49 | 122
  Grade 3 pain | 0 | 0 | 0
  Any redness | 57 | 10 | 9
  Grade 3 redness | 3 | 0 | 0
  Any swelling | 23 | 6 | 7
  Grade 3 swelling | 0 | 0 | 0

2. Primary Outcome: Duration of Solicited Local AEs
Description: Duration was defined as number of days with any grade of local symptoms.
Time Frame: Day 0-6
Population: The analysis was performed on Total Vaccinated cohort which included all subjects with the vaccine administration documented and symptom sheet completed only on subjects that reported the specific symptom.
Measure: Median (Full Range); unit: Days
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 159 | 49 | 122
Days
  Ecchymosis: number analyzed (Participants) | 2 | 3 | 1
  Ecchymosis | 6.5 [6.0 to 7.0] | 5.0 [3.0 to 5.0] | 2.0 [2.0 to 2.0]
  Pain | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 5.0]
  Redness: number analyzed (Participants) | 57 | 9 | 9
  Redness | 3.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 1.0 [1.0 to 6.0]
  Swelling: number analyzed (Participants) | 23 | 6 | 7
  Swelling | 2.0 [1.0 to 7.0] | 1.5 [1.0 to 5.0] | 1.0 [1.0 to 3.0]

3. Primary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General AEs
Description: Any fever was defined as oral temperature ≥38.0 degree centigrade (°C), grade 3 fever was oral temperature ≥ 39.0°C. For other symptoms, any was defined as occurrence of any general symptom regardless of intensity grade or relationship to the study vaccination, grade 3 was defined as a general symptom that prevented normal activity. Related arthralgia, fatigue, gastrointestinal symptoms, headache, myalgia, shivering and fever were defined as general symptoms assessed by the investigator as causally related to the study vaccination.
Time Frame: Day 0-6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 375 | 392 | 203
Participants
  Any arthralgia | 44 | 20 | 11
  Grade 3 arthralgia | 0 | 0 | 1
  Related arthralgia | 25 | 8 | 9
  Any fatigue | 72 | 37 | 39
  Grade 3 fatigue | 1 | 2 | 2
  Related fatigue | 40 | 17 | 28
  Any gastrointestinal symptoms | 26 | 18 | 9
  Grade 3 gastrointestinal symptoms | 1 | 1 | 0
  Related gastrointestinal symptoms | 11 | 10 | 7
  Any headache | 54 | 38 | 31
  Grade 3 headache | 2 | 2 | 0
  Related headache | 33 | 18 | 21
  Any myalgia | 68 | 33 | 36
  Grade 3 myalgia | 0 | 1 | 1
  Related myalgia | 44 | 16 | 26
  Any shivering | 32 | 16 | 10
  Grade 3 shivering | 1 | 2 | 0
  Related shivering | 21 | 8 | 10
  Any fever | 3 | 1 | 2
  Grade 3 fever | 0 | 0 | 0
  Related fever | 3 | 0 | 2

4. Primary Outcome: Duration of Solicited General AEs
Description: Duration was defined as number of days with any grade of general symptoms.
Time Frame: Day 0-6
Population: as for outcome 2
Measure: Median (Full Range); unit: Days
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 72 | 38 | 39
Days
  Arthralgia: number analyzed (Participants) | 44 | 20 | 11
  Arthralgia | 2.0 [1.0 to 7.0] | 3.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Fatigue: number analyzed (Participants) | 72 | 37 | 39
  Fatigue | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Gastrointestinal symptoms: number analyzed (Participants) | 26 | 18 | 9
  Gastrointestinal symptoms | 2.0 [1.0 to 5.0] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Headache: number analyzed (Participants) | 54 | 38 | 31
  Headache | 1.0 [1.0 to 6.0] | 2.0 [1.0 to 7.0] | 1.0 [1.0 to 5.0]
  Myalgia: number analyzed (Participants) | 68 | 33 | 36
  Myalgia | 2.0 [1.0 to 7.0] | 3.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Shivering: number analyzed (Participants) | 32 | 16 | 10
  Shivering | 1.0 [1.0 to 7.0] | 1.5 [1.0 to 5.0] | 2.0 [1.0 to 5.0]
  Fever: number analyzed (Participants) | 3 | 1 | 1
  Fever | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 3.0 [3.0 to 3.0]

5. Primary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited AEs
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade. Grade 3 was defined as an unsolicited symptom that prevented normal activity. Related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: Day 0-20
Population: The analysis was performed on Total Vaccinated cohort which included all subjects with the vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 375 | 393 | 203
Participants
  Any AE(s) | 45 | 47 | 38
  Grade 3 AE(s) | 3 | 8 | 1
  Related AE(s) | 8 | 5 | 3

6. Primary Outcome: Number of Subjects Reporting Any, Grade 3 and Related AEs With a Medically Attended Visit (MAEs) During Day 0 to Day 20
Description: For each solicited and unsolicited AE the subject experienced, the subject was asked if they had received medical attention defined as hospitalization, an emergency room visit or a visit to or from medical personnel (medical doctor) for any reason. Any was defined as occurrence of any symptom regardless of intensity grade, grade 3 was defined as a symptom that prevented normal activity and related was a general symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: Day 0-20
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 375 | 393 | 203
Participants
  Any MAE(s) | 17 | 22 | 9
  Grade 3 MAE(s) | 3 | 6 | 1
  Related MAE(s) | 0 | 0 | 1

7. Primary Outcome: Number of Subjects Reporting AEs of Specific Interest (AESI) Including Autoimmune Diseases From Day 0 to Day 20
Description: AESI for safety monitoring are a subset of AEs that include both clearly autoimmune diseases and also other inflammatory and/or neurologic disorders which may or may not have an autoimmune etiology. Any was defined as occurrence of any symptom regardless of intensity grade.
Time Frame: Day 0-20
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 375 | 393 | 203
Participants | 0 | 0 | 0

8. Primary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs) From Day 0 to Day 20
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade and related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: Day 0-20
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 375 | 393 | 203
Participants
  Any SAEs | 3 | 4 | 0
  Related SAEs | 0 | 0 | 0

9. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related AEs With a Medically Attended Visit (MAEs) Between Day 21 and Day 179
Description: as for outcome 6
Time Frame: Day 21-179
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 375 | 393 | 203
Participants
  Any MAE(s) | 89 | 111 | 55
  Grade 3 MAE(s) | 22 | 26 | 14
  Related MAE(s) | 0 | 0 | 0

10. Secondary Outcome: Number of Subjects Reporting AEs of Specific Interest (AESI) Including Autoimmune Diseases Between Day 21 and Day 364
Description: AESI for safety monitoring are a subset of AEs that include both clearly autoimmune diseases and also other inflammatory and/or neurologic disorders which may or may not have an autoimmune etiology. Any was defined as occurrence of any symptom regardless of intensity grade, grade 3 was defined as a symptom that prevented normal activity and related was a general symptom assessed by the investigator as causally related to the study vaccination.
Time Frame: Day 21-364.
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 375 | 393 | 203
Participants
  Any AESI | 2 | 0 | 0
  Grade 3 AESI | 0 | 0 | 0
  Related AESI | 0 | 0 | 0

11. Secondary Outcome: Haemagglutination Inhibition (HI) Antibody Titers
Description: Antibody titers were expressed as Geometric mean titres (GMTs) per separate vaccine strain. The vaccine strains included A/Brisbane, A/Uruguay and B/Brisbane antigens.
Time Frame: Day 0-21
Population: Analysis was performed on According-to-Protocol (ATP) Immunogenicity cohort. This cohort included all evaluable subjects for whom data concerning immunogenicity were available.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 368 | 375 | 194
titer
  A/Brisbane strain at Day 0: number analyzed (Participants) | 366 | 374 | 194
  A/Brisbane strain at Day 0 | 28.5 [25.7 to 31.5] | 22.9 [20.7 to 25.3] | 52.8 [44.6 to 62.5]
  A/Brisbane strain at Day 21: number analyzed (Participants) | 367 | 375 | 194
  A/Brisbane strain at Day 21 | 70.8 [64.7 to 77.4] | 51.9 [47.0 to 57.2] | 112.5 [98.4 to 128.5]
  A/Uruguay strain at Day 0: number analyzed (Participants) | 366 | 374 | 194
  A/Uruguay strain at Day 0 | 48.9 [43.5 to 54.8] | 29.2 [25.7 to 33.1] | 29.2 [25.1 to 34.0]
  A/Uruguay strain at Day 21: number analyzed (Participants) | 268 | 375 | 194
  A/Uruguay strain at Day 21 | 331.3 [296.7 to 370.0] | 149.2 [131.1 to 169.9] | 161.7 [137.8 to 189.8]
  B/Brisbane strain at Day 0: number analyzed (Participants) | 366 | 374 | 194
  B/Brisbane strain at Day 0 | 169.1 [153.2 to 186.7] | 157.4 [143.2 to 173.1] | 196.4 [167.3 to 230.5]
  B/Brisbane strain at Day 21 | 576.5 [526.5 to 631.1] | 463.5 [422.0 to 509.1] | 765.2 [682.3 to 858.1]

12. Secondary Outcome: The Number of Subjects Seropositive to HI Antibodies
Description: A seropositive subject was defined as a subject with antibody titer greater than or equal to the cut-off value i.e ≥ 1:10. The vaccine strains included A/Brisbane, A/Uruguay and B/Brisbane antigens.
Time Frame: Day 0-21
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 368 | 375 | 194
Participants
  A/Brisbane strain at Day 0: number analyzed (Participants) | 366 | 374 | 194
  A/Brisbane strain at Day 0 | 336 | 315 | 186
  A/Brisbane strain at Day 21: number analyzed (Participants) | 367 | 375 | 194
  A/Brisbane strain at Day 21 | 364 | 366 | 193
  A/Uruguay strain at Day 0: number analyzed (Participants) | 366 | 374 | 194
  A/Uruguay strain at Day 0 | 344 | 320 | 167
  A/Uruguay strain at Day 21 | 368 | 368 | 191
  B/Brisbane strain at Day 0: number analyzed (Participants) | 366 | 374 | 194
  B/Brisbane strain at Day 0 | 366 | 374 | 192
  B/Brisbane strain at Day 21 | 368 | 375 | 194

13. Secondary Outcome: The Number of Subjects Seroprotected by HI Antibodies
Description: A seroprotected subject was defined as a subject with a serum HI titer ≥ 1:40 that usually is accepted as indicating protection. The vaccine strains included A/Brisbane, A/Uruguay and B/Brisbane antigens.
Time Frame: Day 0-21
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 368 | 375 | 194
Participants
  A/Brisbane strain at Day 0: number analyzed (Participants) | 366 | 374 | 194
  A/Brisbane strain at Day 0 | 171 | 142 | 137
  A/Brisbane strain at Day 21: number analyzed (Participants) | 367 | 375 | 194
  A/Brisbane strain at Day 21 | 314 | 276 | 179
  A/Uruguay strain at Day 0: number analyzed (Participants) | 366 | 374 | 194
  A/Uruguay strain at Day 0 | 247 | 178 | 102
  A/Uruguay strain at Day 21 | 361 | 341 | 181
  B/Brisbane strain at Day 0: number analyzed (Participants) | 366 | 374 | 194
  B/Brisbane strain at Day 0 | 359 | 363 | 186
  B/Brisbane strain at Day 21 | 368 | 375 | 194

14. Secondary Outcome: The Number of Subjects Seroconverted to HI Antibodies
Description: A seroconverted subject was defined as a subject who had either a pre-vaccination titer < 1:10 and a post-vaccination titer ≥ 1:40 or a pre-vaccination titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer. The vaccine strains included A/Brisbane, A/Uruguay and B/Brisbane antigens.
Time Frame: At Day 21
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 366 | 374 | 194
Participants
  A/Brisbane strain | 107 | 94 | 54
  A/Uruguay strain | 285 | 228 | 124
  B/Brisbane strain | 168 | 140 | 104

15. Secondary Outcome: HI Antibody Seroconversion Factors (SCF)
Description: SCF was defined as the fold increase in serum HI GMTs post-vaccination compared to Day 0. The vaccine strains included A/Brisbane, A/Uruguay and B/Brisbane antigens.
Time Frame: At Day 21
Population: Analysis was performed on According-to-Protocol (ATP) immunogenicity cohort . The cohort included all evaluable subjects for whom data concerning immunogenicity at were available.
Measure: Mean (95% Confidence Interval); unit: fold increase
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 366 | 374 | 194
fold increase
  A/Brisbane strain | 2.5 [2.3 to 2.7] | 2.3 [2.1 to 2.5] | 2.1 [1.9 to 2.4]
  A/Uruguay strain | 6.8 [6.1 to 7.5] | 5.1 [4.6 to 5.7] | 5.5 [4.7 to 6.5]
  B/Brisbane strain | 3.4 [3.1 to 3.7] | 2.9 [2.7 to 3.2] | 3.9 [3.3 to 4.5]

16. Secondary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs) From Day 21 to Day 364
Description: as for outcome 8
Time Frame: Day 21-364
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Number analyzed (Participants) | 375 | 393 | 203
Participants
  Any SAE(s) | 40 | 43 | 4
  Related SAE(s) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events were assessed from Day 0 to 20 and from Day 21 to 364. Systematically assessed frequent adverse events (AEs) and non-systematically assessed frequent AEs were assessed during 7 day and 21 day post-vaccination period respectively.
Description: For the frequent adverse events, the number of participants at risk included those from Total Vaccinated Cohort who had the symptom sheet completed.
Arm/Group | New Generation Influenza Vaccine GSK2186877A Group | Fluarix Elderly Group | Fluarix Young Group
Serious Adverse Events (participants affected / at risk) | 40/375 | 43/393 | 4/203
Other Adverse Events (participants affected / at risk) | 218/375 | 109/393 | 133/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | New Generation Influenza Vaccine GSK2186877A Group (N=375) | Fluarix Elderly Group (N=393) | Fluarix Young Group (N=203)
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 — SAE was assessed from Day 0 to Day 20
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — SAE was assessed from Day 0 to Day 20
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 — SAE was assessed from Day 0 to Day 20
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 — SAE was assessed from Day 0 to Day 20
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 — SAE was assessed from Day 0 to Day 20
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 — SAE was assessed from Day 0 to Day 20
Urosepsis (Infections and infestations) | 0 | 1 | 0 — SAE was assessed from Day 0 to Day 20
Hip fracture (Injury, poisoning and procedural complications) | 3 | 1 | 0 — SAE was assessed from Day 21-364
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 — SAE was assessed from Day 21-364
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 — SAE was assessed from Day 21-364
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 — SAE was assessed from Day 21-364
Urosepsis (Infections and infestations) | 1 | 1 | 0 — SAE was assessed from Day 21-364
Coronary artery occlusion (Cardiac disorders) | 1 | 1 | 0 — SAE was assessed from Day 21-364
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 — SAE was assessed from Day 21-364
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 — SAE was assessed from Day 21-364
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — SAE was assessed from Day 21-364
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — SAE was assessed from Day 21-364
Pneumonia staphylococcal (Infections and infestations) | 1 | 0 | 0 — SAE was assessed from Day 21-364
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2 | 0 — SAE was assessed from Day 21-364
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 0 — SAE was assessed from Day 21-364
Myocardial infarction (Cardiac disorders) | 1 | 3 | 0 — SAE was assessed from Day 21-364
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 — SAE was assessed from Day 21-364
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 — SAE was assessed from Day 21-364
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 0 — SAE was assessed from Day 21-364
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 — SAE was assessed from Day 21-364
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 — SAE was assessed from Day 21-364
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 1 | 0 — SAE was assessed from Day 21-364
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 0 — SAE was assessed from Day 21-364
Diverticulitis (Infections and infestations) | 1 | 0 | 0 — SAE was assessed from Day 21-364
Chest pain (General disorders) | 1 | 2 | 0 — SAE was assessed from Day 21-364
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 — SAE was assessed from Day 21-364
Pneumonia (Infections and infestations) | 3 | 3 | 0 — SAE was assessed from Day 21-364
Fatigue (General disorders) | 1 | 0 | 0 — SAE was assessed from Day 21-364
Angina pectoris (Cardiac disorders) | 1 | 1 | 0 — SAE was assessed from Day 21-364
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 — SAE was assessed from Day 21-364
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 — SAE was assessed from Day 21-364
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 — SAE was assessed from Day 21-364
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 — SAE was assessed from Day 21-364
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 — SAE was assessed from Day 21-364
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 — SAE was assessed from Day 21-364
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 — SAE was assessed from Day 21-364
Adverse drug reaction (General disorders) | 1 | 0 | 0 — SAE was assessed from Day 21-364
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 — SAE was assessed from Day 21-364
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 — SAE was assessed from Day 21-364
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 — SAE was assessed from Day 21-364
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 — SAE was assessed from Day 21-364
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0 — SAE was assessed from Day 21-364
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 — SAE was assessed from Day 21-364
Volvulus (Gastrointestinal disorders) | 1 | 0 | 0 — SAE was assessed from Day 21-364
Viral infection (Infections and infestations) | 1 | 0 | 0 — SAE was assessed from Day 21-364
Death (General disorders) | 1 | 0 | 0 — SAE was assessed from Day 21-364
Bronchitis (Infections and infestations) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Cystocele (Reproductive system and breast disorders) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Haemorrhagic stroke (Nervous system disorders) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Left ventricular failure (Cardiac disorders) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Enterocolitis infectious (Infections and infestations) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Lymphatic fistula (Vascular disorders) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Wound infection (Infections and infestations) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Factor XIII deficiency (Congenital, familial and genetic disorders) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Herpes zoster (Infections and infestations) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 — SAE was assessed from Day 21-364
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Stress cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Aesthesioneuroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Sepsis (Infections and infestations) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Chest discomfort (General disorders) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Femoral arterial stenosis (Vascular disorders) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Appendicitis (Infections and infestations) | 0 | 1 | 2 — SAE was assessed from Day 21-364
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 — SAE was assessed from Day 21-364
Dizziness (Nervous system disorders) | 0 | 0 | 1 — SAE was assessed from Day 21-364
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 — SAE was assessed from Day 21-364
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | New Generation Influenza Vaccine GSK2186877A Group (N=375) | Fluarix Elderly Group (N=393) | Fluarix Young Group (N=203)
Pain (General disorders) | 159 | 49 | 122
Redness (General disorders) | 57 | 10 | 9
Swelling (General disorders) | 23 | 6 | 7
Arthralgia (General disorders) | 44 | 20 | 11
Fatigue (General disorders) | 72 | 37 | 39
Gastrointestinal symptoms (General disorders) | 26 | 18 | 9
Headache (General disorders) | 54 | 38 | 31
Myalgia (General disorders) | 68 | 33 | 36
Shivering (General disorders) | 32 | 16 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.